CLINICAL TRIAL: NCT00261989
Title: The Retrospective Analysis of Presenting Pulse Oximetry Readings and Hourly Variation in Oximetry Readings in Patients With Known Congenital Heart Disease
Brief Title: Pulse Oximetry Readings and Hourly Variation in Oximetry Readings With CHD
Status: Terminated | Type: Observational
Why Stopped: data insignificant, study terminated
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-198
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-09

CONDITIONS: Congenital Disorders
Keywords: pulse oximetry readings; pediatrics; cardiac; congenital heart disease
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heart Defects, Congenital

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to describe the presenting pulse oximetry reading in patients who have a known lesion which will cause them to have a low presenting oximetry reading. The study hypothesis is that there is a low presenting pulse oximetry in patients with congenital heart disease and that there will be no significant variation in the hourly variation in oximetry readings in these patients.

DETAILED DESCRIPTION:
Congenital heart disease is a relatively common disease seen in 8/1,000 live births. Many of these diseases are associated with hypoxemia. Hypoxemia results from the mixing of pulmonary and systemic blood or from the mixing of parallel circulations as seen in transposition of the great vessels. Pulse oximetry can be used to measure hypoxemia. Pulse oximetry estimates oxygen saturation by measuring absorption of light in human tissue beds. The amount of light absorption varies depending on the amount of deoxygenated blood in the tissue measured. Measuring the changes in light absorption allows for an estimation of arterial oxygen saturation and therefore the amount of hypoxemia. Most manufacturers claim a confidence interval of 4% for their oximeters. There have been a few studies recently describing the presenting pulse oximetry of known congenital heart disease. However, these were small studies with a small sample size of patients. Moreover, there is no literature describing the hourly variation in pulse oximetry among know congenital heart disease patients.

We hypothesize that there is a low presenting pulse oximetry in patients with congenital heart disease and that there will be no significant variation in the hourly variation in oximetry readings in these patients.

This is a retrospective chart review examining the presenting pulse oximetry of patients with known cyanotic heart lesions. The treatment group will be untreated patients with known lesions. All charts of children presenting to Sibley Heart Center with known cyanotic heart lesions from January 1, 2004 to December 31, 2004 will be reviewed.

The aim of the study is to describe the presenting pulse oximetry reading in patients who have a known lesion which will cause them to have a low oximetry reading. The following information will be collected from the charts:

* Presenting pulse oximetry
* Heart lesion

The second aim will be to characterize the hourly variation in pulse oximetry from these patients. The following information will be collected:

* Hourly pulse oximetry readings
* Heart lesion
* Clinical course

ELIGIBILITY:
Inclusion Criteria:

* congenital heart lesion
* presenting to Sibley Heart Center
* initial visit between Jan. 1, 2004 and Dec. 31, 2004

Exclusion Criteria:

* those who do not meet inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: retro chart review
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2005-11; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Mahle, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States